CLINICAL TRIAL: NCT06386848
Title: Strategy to Adapt Botulinum Toxin Doses in Dystonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Solène FRISMAND, Dr Kryllof-Frismand Solène, Central Hospital, Nancy, France
Other Study IDs: 2023PI187
Record Dates: First submitted 2024-01-18; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-01

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Botulinum Toxins; Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Botulinum toxin — Botulinum toxin doses injected in dystonia
  Other Names: onabotulinumtoxinA, abobotulinumtoxinA, incobotulinumtoxinA

SUMMARY:
The study is designed to observ and collect the doses of botulinum toxin injected in dystonia in different centres to compare the initial dose and the dose recommended.

We we ll study the increase of the dose injected over the time, the side effects...

The hypothesis is that we inject smaller doses than we could regarding the recommandations

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old followed for dystonia and treated with botulinum toxin

Exclusion Criteria:

* first dose of botulinum toxin not available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years diagnosed with dystonia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
First dose of botulinum toxin injected, U | 30 years
  dose injected in U

SECONDARY OUTCOMES:
Effective dose of botulinum toxin | 30 years
  dose injected in U
Side effects | 30 years
  diplopia, ptosis and others